CLINICAL TRIAL: NCT05170516
Title: The Effect of Saline Irrigation at Different Temperatures on Pain, Edema, and Trismus After Impacted Third Molar Surgery: A Prospective, Randomized, Split-Mouth, Clinical Trial
Brief Title: The Effect of Saline Irrigation at Different Temperatures on Pain, Edema, and Trismus After Impacted Third Molar Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Fatma Gülfeşan Çanakçi, Assistant Professor, Trakya University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TrakyaU 2018
Record Dates: First submitted 2021-12-21; First posted 2021-12-28 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-01

CONDITIONS: Impacted Third Molar Tooth
Keywords: Cooled irrigation; Impacted third molar; Postoperative morbidity; Cooled saline

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental Group A (Experimental): In experimental group A, 4°C saline irrigation was used for removal of the bone surrounding the right or left third molars.
  Interventions: Procedure: 4 °C colled saline irrigation
- Experimental Group B (Experimental): In experimental group B, 10°C saline irrigation was used for removal of the bone surrounding the right or left third molars.
  Interventions: Procedure: 10 °C cooled saline irrigation
- Control Group A (Active Comparator): In control group A, room temperature saline was used for the other side extractions of patients whose impacted tooth was extracted under 4 °C saline irrigation on one side.
  Interventions: Procedure: Room temperature saline irrigation
- Control Group B (Active Comparator): In control group B, room temperature saline was used for the other side extractions of patients whose impacted tooth was extracted under 10 °C saline irrigation on one side.
  Interventions: Procedure: Room temperature saline irrigation

INTERVENTIONS:
Procedure: 4 °C colled saline irrigation — In Experimental Group A , 4 °C colled saline irrigation was used during impacted third molar surgery
  Arms: Experimental Group A
Procedure: 10 °C cooled saline irrigation — Experimental Group B, 10°C colled saline irrigation was used during impacted third molar surgery.
  Arms: Experimental Group B
Procedure: Room temperature saline irrigation — In Control Group A and B, salin irrigation at room temperature was used during impacted third molar surgery.
  Arms: Control Group A; Control Group B

SUMMARY:
Third molar surgery is one of the most common procedures in oral surgery and the most common postoperative complications are swelling, pain, and trismus. This study aims to evaluate the postoperative morbidity (pain, swelling, and trismus) in third molar surgery performed using different degrees of cooled and room temperature irrigation solutions.

DETAILED DESCRIPTION:
This single-blind, single- centre, split-mouth, superiority randomized prospective clinical trial was approved by The Ethics Committee of Trakya University, Medical Sciences (Decision no: 13/10). The sample size calculation based on data obtained from a previous study indicated that 48 patients would be sufficient per group (80% power and 5% significance level).

Adult patients (18 - 59 years of age) referred to the Trakya University, Faculty of Dentistry, Department of Oral and Maxillofacial Surgery between September 2018 and December 2020 were examined clinically and radiographically.

Inclusion criteria:

1. Patients who fit the requirements of the study such as attending follow up sessions and signing the informed consent.
2. Patients who had bilateral asymptomatic vertical third molar teeth with impaction of class I, level C (21).
3. Patients who had no significant medical diseases or use of drugs, were not pregnant, had no allergy, and did not smoke.

A patient was excluded if any of the following conditions were observed:

1. Patients who have a complicating systemic disease (ASA: 3- 6).
2. Patients who have second molars with severe periodontal defect or deep periodontal pocket (probing depth >4mm)
3. Patients who have a poor oral hygiene
4. Patients who have history of having taken analgesics 12 h or antibiotics 1 month before.

Fourty eight patients were randomly allocated to two groups (Group A and B)(n =24). For randomization, a dentist blinded to the study took a sealed envelope from the bag, which contained group codes. Bilateral impacted third molars (a total of 96 teeth) were extracted from each patient in 2 different operation time. The second operation that was performed at least 21 days after the first ones to return the variables to preoperative values. Each patient had an experimental (one side with 4°C or 10°C saline irrigation) and control (the other side with 25°C saline irrigation ) group impacted third molars.

All procedures were completed by a single operator who had ten years of experience. Inferior alveolar nerve, lingual and buccal nerve blocks were performed using a local anesthetic containing 0.006 mg/ml adrenaline hydrochloride and 40 mg/ml articaine hydrochloride (2 ml Ultracaine® D-S Ampul, Sanofi Aventis). The flap was released with a triangular incision. Osteotomies were made with a 1.6 mm round bur attached to a surgical high-speed handpiece (W&H Implantmed, W&H, St Albans, UK) at 20000 rpm under saline irrigation at the temperature determined according to the groups.

During operations, the temperatures of the salines were verified with a non-contact thermometer (Omron Gentle Temp 720 MC, Omron Healthcare Co., Ltd., Kyoto, Japan) every 30 seconds. When temperature changes were detected, the correct temperature was achieved with the addition of cooled irrigation. After tooth extraction flap was sutured with a 3.0 silk suture which was removed 7 days after the surgery. The operation time was determined as the time between the first incision and the last suture and recorded.

Biting a gauze pack for 30 minutes, an ice pack compression (5 minutes on and 5 minutes off) for 6 hours, and having a soft and cold diet for 24 hours were recommended. Amoxicillin 500 mg 3 times/day for 5 days and 0.12% chlorhexidine digluconate mouthwash 3 times/day for 7 days were prescribed. The patients were also advised to take paracetamol 500 mg as required.

Assessment of postoperative pain before participation, all patients had read and signed an informed consent form. All patients were given a pain form to report the level of postoperative pain. Before the beginning of treatment, the clinician filled in an example of a pain report with each patient to confirm that they understood the instructions. Postoperative pain was evaluated by the Visual Analogue Scale (VAS) from "0" (as no pain) to "10" (as the most severe pain experienced) for postoperative 7 days. And also patients were asked to record the number of analgesics they used in 1 day for 7 days. Patients were not aware of the side and the type of cooled irrigation in order not to affect VAS scores and the total number of analgesics.

Postoperative measurements were made by a single surgeon blinded to operative procedures. Patients were recalled on the 24th and 72nd hours and 7th days postoperatively, and trismus and facial swelling measurements were made.

The level of facial swelling was determined by a method described by Üstün et. al. (22). To assess facial swelling, three measurements between 5 reference points were performed with a flexible ruler: tragus to soft tissue pogonion, lateral corner of the eye to the angle of the mandible, and tragus to the outer corner of the mouth. The sum of the 3 measurements was calculated preoperatively and repeated on postoperative days 1, 3, and 7. The difference between each postoperative measurement and the preoperative measurement was determined as the value for facial swelling.

Trismus was assessed by measuring the distance between the mesial incisal corners of the right upper and lower central teeth when the patient had maximum mouth opening on postoperative 1, 3, 7 days. The difference between each postoperative measurement and the preoperative measurement indicated the trismus for that day.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers over the age of 18
* Patients who had no significant medical diseases or use of drugs, were not pregnant, had no allergy, and did not smoke.
* Patients who had bilateral asymptomatic vertical third molar teeth with impaction of class I, level C according to Pell and Gregory Classification, and no history of recent antibiotic or anti-inflammatory treatment.

Exclusion Criteria:

* Patients who had symptomatic impacted third molars.
* Patients who had a medical history described above.
* Patients under the age of 18.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-09-15 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Change in trismus | 7 days
  Trismus was assessed by measuring the distance between the mesial incisal corners of the right upper and lower central teeth when the patient had maximum mouth opening. The difference between each postoperative measurement and the preoperative measurement indicated the trismus for that day.
Change in Facial Swelling | 7 days
  three measurements between 5 reference points were performed with a flexible ruler: tragus to soft tissue pogonion, lateral corner of the eye to the angle of the mandible, and tragus to the outer corner of the mouth. The sum of the 3 measurements was calculated preoperatively and repeated.The difference between each postoperative measurement and the preoperative measurement was determined as the value for facial swelling.
Change in pain | 7 days
  Postoperative pain was evaluated by the Visual Analogue Scale (VAS) from "0" (as no pain) to "10" (as the most severe pain experienced).

SECONDARY OUTCOMES:
Change in the number of analgesic | 7 days
  patients were asked to record the number of analgesics they used.

CONTACTS AND LOCATIONS:
Overall Officials: F. Gülfeşan Çanakçi, Study Director — Trakya University, Faculty of Dentistry
Locations (1):
- Trakya University, Edirne, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No